CLINICAL TRIAL: NCT07280208
Title: Impact of Discharge Teach-Back Education on Heart Failure Patients' Knowledge/Self-Care Behaviors and 30-Day Readmissions
Brief Title: Teach-Back Discharge Education to Improve Self-Care and Reduce 30-Day Readmissions in Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Responsible Party: Principal Investigator, Sara Bierschenk, Principal Investigator, Nova Southeastern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025-398
Record Dates: First submitted 2025-11-29; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure; Heart Failure Hospitalization; Readmission, Hospital
Keywords: heart failure; hospital readmission; patient education; teach-back method; self-care; health literacy; discharge planning; transitional care; evidence-based practice; nursing intervention; quality improvement; systolic heart failure; medication adherence; symptom monitoring; lifestyle modification
MeSH Terms: conditions — Heart Failure; Heart Failure, Systolic; Medication Adherence

STUDY DESIGN:
Intervention Model Description: All participants receive the same intervention: structured discharge education using the teach-back method.
  There is no control group or comparison between multiple interventions. The study uses a pre-test/post-test design within a single group to evaluate changes in self-care behaviors and readmission rates.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Teach-Back Education Intervention (Experimental): Participants in this arm will receive a structured discharge education session using the teach-back method. The session will be delivered in person at hospital discharge and will cover key heart failure self-care behaviors, including medication adherence, symptom monitoring, fluid restriction, and dietary modifications. Participants will be asked to restate instructions in their own words to confirm understanding. Printed educational materials from the American Heart Association will also be provided.
  Interventions: Behavioral: Teach-Back Discharge Education

INTERVENTIONS:
Behavioral: Teach-Back Discharge Education — A structured, 30-minute discharge education session delivered in person using the teach-back method. Participants are asked to restate instructions in their own words to confirm understanding. The session covers key heart failure self-care behaviors including medication adherence, symptom monitoring, fluid restriction, and dietary modifications. Printed educational materials from the American Heart Association are also provided.

SUMMARY:
This study aims to improve how patients with heart failure understand and manage their condition after leaving the hospital. Many heart failure patients are readmitted within 30 days due to confusion about their discharge instructions and difficulty following self-care routines. The study will test whether a structured discharge education session using the "teach-back" method-where patients repeat instructions in their own words-can help improve their knowledge and self-care behaviors. The goal is to reduce hospital readmissions and help patients feel more confident managing their heart failure at home.

DETAILED DESCRIPTION:
Heart failure is a chronic and progressive condition affecting millions of adults in the United States. Despite advances in treatment, nearly one in four patients are readmitted to the hospital within 30 days of discharge, often due to poor understanding of discharge instructions and inadequate self-care. These readmissions contribute to worse health outcomes and increased healthcare costs.

This study evaluates the effectiveness of a structured discharge education intervention using the teach-back method. The teach-back method is a communication technique in which patients are asked to repeat discharge instructions in their own words. This approach helps confirm understanding, reinforce learning, and promote active engagement in self-care.

The study uses a quasi-experimental, pre-test/post-test design to assess changes in patients' knowledge and self-care behaviors before and after the intervention. Participants are adults hospitalized with systolic heart failure (LVEF ≤ 40%) who meet specific clinical criteria. Each participant receives a 30-minute individualized education session at discharge, covering key self-care topics such as medication adherence, symptom monitoring, fluid restriction, and dietary modifications. Printed educational materials from the American Heart Association are also provided.

To measure outcomes, participants complete the European Heart Failure Self-care Behavior Scale (EHFScB-9) before and after the intervention. Thirty-day readmission data are collected through a retrospective review of hospital records. The study aims to determine whether teach-back education improves self-care behaviors and reduces 30-day readmission rates.

This project has been reviewed and exempted by the Nova Southeastern University Institutional Review Board under Exempt Category 2. It aligns with national goals to improve patient education, reduce preventable readmissions, and enhance the quality of care for individuals with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Diagnosed with systolic heart failure with a left ventricular ejection fraction (LVEF) ≤ 40%
* Classified as New York Heart Association (NYHA) Class II, III, or IV
* Categorized as American College of Cardiology/American Heart Association (ACC/AHA) Stage C or D
* Currently hospitalized at the project site
* Able to read and understand English at an 8th grade reading level
* Have access to a smartphone or tablet capable of scanning QR codes and connecting to the internet
* Provide voluntary informed consent via the REDCap platform

Exclusion Criteria:

* Cognitive impairment
* Non-English speaking
* Unwilling to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2025-09-11 (Actual); Primary Completion 2025-10-11 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Change in Heart Failure Self-Care Behaviors | Baseline (pre-intervention) and immediately post-discharge (post-intervention)
  Assessed using the European Heart Failure Self-care Behavior Scale (EHFScB-9), a validated 9-item questionnaire. Each item is rated on a 5-point Likert scale from 1 ("completely agree") to 5 ("do not agree at all").
  Total scores range from 9 to 45, with lower scores indicating better self-care behaviors.
  The outcome will be measured as the change in total score from pre- to post-intervention.
Change in Heart Failure Self-Care Behaviors | Baseline (pre-intervention) and immediately post-discharge (post-intervention)
  Assessed using the European Heart Failure Self-care Behavior Scale (EHFScB-9), a validated 9-item questionnaire measuring frequency and consistency of self-care practices such as daily weight monitoring, medication adherence, and symptom recognition. Each item is rated on a 5-point Likert scale from 1 ("completely agree") to 5 ("do not agree at all").
  Total scores range from 9 to 45, with lower scores indicating better self-care behaviors.
  The outcome will be measured as the change in total score from pre- to post-intervention.

SECONDARY OUTCOMES:
30-Day Heart Failure Readmission Rate | 30 days post-discharge
  Readmission status will be determined by reviewing hospital records to identify whether participants were readmitted for heart failure within 30 days of discharge.
  Participants will be classified as readmitted (Yes) or not readmitted (No) based on whether a heart failure-related hospitalization occurred within the 30-day period.
  The outcome will be reported as the percentage of participants readmitted within 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Waters, Ph.D., MSN, MBA, RN, CNE-BC, Study Chair — Nova Southeastern University, Ron and Kathy Assaf College of Nursing
Locations (1):
- HCA Florida JFK Hospital, Atlantis, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared for this study. The data collected will be used solely for the purposes of evaluating the effectiveness of the discharge teach-back education intervention on heart failure self-care behaviors and 30-day readmissions. All data will be stored securely and managed in compliance with HIPAA and IRB regulations. Due to the sensitive nature of health information and the limited scope of the study, there is no plan to make IPD publicly available.